CLINICAL TRIAL: NCT02835690
Title: An Open-label, Randomized Phase I Study Investigating Safety, Tolerability, Pharmacokinetics, and Efficacy of Pembrolizumab (MK-3475) in Chinese Subjects With Non-Small-Cell Lung Cancer
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Pembrolizumab (MK-3475) in Chinese Participants With Non-Small-Cell Lung Cancer (MK-3475-032/KEYNOTE-032)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-032; MK-3475-032 (Other: Merck Protocol Number); KEYNOTE-032 (Other: Merck)
Record Dates: First submitted 2016-06-29; First posted 2016-07-18 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-09

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pembrolizumab 2 mg/kg (Experimental): Participants will receive pembrolizumab 2 mg/kg administered intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab 10 mg/kg (Experimental): Participants will receive pembrolizumab 10 mg/kg administered IV Q3W for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab 200 mg Fixed Dose (Experimental): Participants will receive pembrolizumab 200 mg fixed dose administered IV Q3W for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and efficacy of three doses of pembrolizumab (MK-3475) in adult Chinese participants with locally advanced or metastatic non-small-cell lung cancer (NSCLC).

Cycle 1 is 28 days long; subsequent cycles are 21 days long.

ELIGIBILITY:
Inclusion Criteria:

* Is of the Chinese race (i.e., Chinese descent born in China) and has a Chinese home address.
* Has a life expectancy of at least 3 months.
* Has histologically-/cytologically-confirmed, advanced unresectable NSCLC and has measurable disease based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by the site.
* Has failed established standard medical anti-cancer therapies or has been intolerant to such therapy, or in the opinion of the investigator have been considered ineligible for any form of standard therapy on medical grounds.
* Has a score of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status within 3 days prior to the first dose of study drug.
* Has adequate organ function.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
* Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* Has had chemotherapy, radioactive, or biological cancer therapy within 4 weeks prior to the first dose of study therapy pembrolizumab, or who has not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the AEs due to cancer therapeutics administered more than 4 weeks earlier.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* Is expected to require any other form of antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC).
* Has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication.
* Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the participant has undergone potentially curative therapy with no evidence of that disease for 5 years.
* Has known central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Had prior treatment targeting PD-1: PD-L1 axis or cytotoxic T-lymphocyte-associated protein, or was previously randomized in any pembrolizumab study. Examples of such agents include (but are not limited to): Nivolumab (BMS-936558, MDX-1106 or ONO-4538); Pidilizumab (CT-011); AMP-224; BMS-936559 (MDX-1105); MPDL3280A (RG7446); and MEDI4736.
* Has an active infection requiring systematic therapy.
* Is positive for Human Immunodeficiency Virus.
* Has known active Hepatitis B or C.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received or will receive a live vaccine within 30 days prior to the first administration of study drug.
* Is at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Is pregnant or breastfeeding, or expecting to conceive or father a child within the projected duration of the study, starting with the screening visit (Visit 1) through 120 days after the last dose of pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ma Y, Fang W, Zhang Y, Yang Y, Hong S, Zhao Y, Xie S, Ge J, Zhou H, Zhao H, Zhang L. KEYNOTE-032: A Randomized Phase I Study of Pembrolizumab in Chinese Patients with Advanced Non-Small Cell Lung Cancer. Oncologist. 2020 Aug;25(8):650-e1145. doi: 10.1634/theoncologist.2020-0067. Epub 2020 Mar 5. PMID 32134163
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 44 participants randomized, 42 received treatment. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab 2 mg/kg: Participants received pembrolizumab 2 mg/kg administered intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Pembrolizumab 10 mg/kg: Participants received pembrolizumab 10 mg/kg administered IV Q3W for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Pembrolizumab 200 mg Fixed Dose: Participants received pembrolizumab 200 mg fixed dose administered IV Q3W for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Period: Overall Study
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Started | 14 | 15 | 15
Received First Course of Pembrolizumab | 14 | 13 | 15
Received Second Course of Pembrolizumab | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 14 | 15 | 15
Not completed — Death | 12 | 11 | 13
Not completed — Transferred to Extension Study | 2 | 2 | 1
Not completed — Did Not Continue on Extension Study | 0 | 0 | 1
Not completed — Not Treated | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants that received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose | Total
Number analyzed (Participants) | 14 | 13 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.5) | 56.2 (11.5) | 56.7 (8.8) | 55.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 9 | 9 | 9 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 13 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 14 | 13 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to be a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who experienced at least one AE was reported per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab 2 mg/kg: Participants receive pembrolizumab 2 mg/kg administered intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days.
- Pembrolizumab 10 mg/kg: Participants receive pembrolizumab 10 mg/kg administered IV Q3W for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days.
- Pembrolizumab 200 mg Fixed Dose: Participants receive pembrolizumab 200 mg fixed dose administered IV Q3W for up to 35 administrations. Cycle 1 is 28 days and subsequent cycles are 21 days.
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Participants | 14 | 13 | 14

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to be a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who discontinued study treatment due to an AE was reported per protocol for the first course of treatment.
Time Frame: Up to ~12 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Participants | 0 | 1 | 3

3. Primary Outcome: Single Dose PK: Area Under the Plasma Concentration Curve From 0-28 Days (AUC[0-28 Days]) of Pembrolizumab
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected pre-dose and post-dose at multiple time points up to 28 days during cycle 1 to estimate AUC(0-28 days) following single dose administration for the first course of treatment.
Time Frame: Cycle 1 Day 1: pre-dose [-1 to 0 hour] and post-dose at 0 [up to 0.5], 6 [±0.5], 24, 48, 168, 336, and 504 [±2 for 24 to 504] hours after completion of pembrolizumab infusion. Cycle 1= 28 days
Population: All randomized participants who received a pembrolizumab dose, with available pharmacokinetic (PK) data, and who did not have any protocol deviation interfering with PK.
Measure: Geometric Mean (95% Confidence Interval); unit: μg•day/mL
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
μg•day/mL | 437.10 [388.94 to 491.22] | 1979.62 [1737.75 to 2255.15] | 637.22 [569.89 to 712.51]

4. Primary Outcome: Single-Dose PK: Maximum Plasma Concentration (Cmax) of Pembrolizumab
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected pre-dose and post-dose at multiple time points up to 28 days during cycle 1 to estimate Cmax following single dose administration for the first course of treatment.
Time Frame: as for outcome 3
Population: All randomized participants who received a pembrolizumab dose, with available PK data, and who did not have any protocol deviation interfering with PK.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
μg/mL | 50.62 [42.34 to 60.52] | 213.12 [191.45 to 237.25] | 76.21 [63.59 to 91.32]

5. Primary Outcome: Single Dose PK: Time to Cmax (Tmax) of Pembrolizumab
Description: Tmax was defined as the time required post dosing to reach a maximum plasma concentration of pembrolizumab. Blood samples were collected pre-dose and post-dose at multiple time points up to 28 days at cycle 1 to estimate Tmax following single dose administration for the first course of treatment.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: day
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
day | 0.06 [0.03 to 2.02] | 0.05 [0.02 to 0.27] | 0.04 [0.02 to 0.27]

6. Primary Outcome: Single Dose PK: Apparent Terminal Half-Life (t1/2) of Pembrolizumab
Description: t½ was defined as the time required to divide the pembrolizumab plasma concentration by two after reaching pseudo-equilibrium, following a single dose of pembrolizumab. Blood samples were collected pre-dose and post-dose at multiple time points up to 28 days at cycle 1 to estimate t½ following single dose administration for the first course of treatment.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: Day
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Day | 14.10 [9.56 to 31.60] | 16.00 [10.50 to 23.80] | 12.70 [4.15 to 24.50]

7. Primary Outcome: Multiple Dose PK: Trough Plasma Concentration (Ctrough) of Pembrolizumab
Description: Ctrough was defined as the minimum concentration that occurred immediately prior to the administration of pembrolizumab in Cycle 8. Blood samples were collected pre-dose at Cycle 8 to estimate Ctrough following multiple dose administrations of pembrolizumab for the first course of treatment.
Time Frame: Cycle 8 Day 1: pre-dose [-1 to 0 hour]. (Cycle 1 = 28 days, Cycles 2-8 = 21 days).
Population: All randomized participants who received a pembrolizumab dose, had available Ctrough data, and who did not have any protocol deviation interfering with PK.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 8 | 5 | 5
μg/mL | 21.53 [15.76 to 29.41] | 78.35 [56.09 to 109.45] | 25.46 [17.70 to 36.63]

8. Primary Outcome: Multiple Dose PK: AUC(0-21 Days) of Pembrolizumab at Steady State
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time at steady state following multiple doses. Blood samples were collected pre-dose and post-dose at multiple time points up to 21 days during cycle 8 to assess AUC(0-21 days) at steady state for the first course of treatment.
Time Frame: Cycle 8 Day 1: pre-dose [-1 to 0 hour] and post-dose at 0 [up to 0.5], 6 [up to 0.5], 24, 48, 168, 336, and 504 [±2 for 24 to 504] hours after completion of pembrolizumab infusion. Cycle 8 up to 175 days (Cycle 1 = 28 days, Cycles 2-8 = 21 days).
Population: All randomized participants who received a pembrolizumab dose, had available AUC(0-21 days) data, and who did not have any protocol deviation interfering with PK.
Measure: Geometric Mean (95% Confidence Interval); unit: μg•day/mL
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 7 | 5 | 4
μg•day/mL | 730.94 [627.38 to 851.60] | 2819.19 [2009.36 to 3955.43] | 930.99 [724.37 to 1196.56]

9. Primary Outcome: Multiple Dose PK: Cmax of Pembrolizumab at Steady State
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma at steady state following multiple doses. Blood samples were collected pre-dose and post-dose at multiple time points up to 21 days during cycle 8 to assess Cmax assessment at steady state for the first course of treatment.
Time Frame: as for outcome 8
Population: All randomized participants who received a pembrolizumab dose, had available Cmax data, and who did not have any protocol deviation interfering with PK.
Measure: Geometric Mean (95% Confidence Interval); unit: g/mL
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 8 | 5 | 5
g/mL | 66.67 [56.90 to 78.10] | 268.59 [217.81 to 331.21] | 92.22 [81.66 to 104.16]

10. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Central Radiologists' Review
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: disappearance of all lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions, without evidence of progression based on non-target or new lesions) as assessed by central radiologists' review per RECIST 1.1 which is modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a confirmed CR or PR per RECIST 1.1 as assessed by central radiologists' review was reported for each arm per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment and with measurable disease at baseline as assessed by central radiology review.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Percentage of participants | 0.0 [0.0 to 23.2] | 23.1 [5.0 to 53.8] | 20.0 [4.3 to 48.1]

11. Secondary Outcome: ORR Per Immune-related RECIST (irRECIST) as Assessed by Central Radiologists' Review
Description: ORR was defined as the percentage of participants who had confirmed responses assessed using RECIST 1.1 before PD or an immune-related Complete Response (irCR: Disappearance of all target lesions and non-target) or an immune-related Partial Response (irPR: At least a 30% decrease in the sum of diameters of target lesions, stability of non-target lesions no new lesions) after a single PD per irRECIST as assessed by central radiologists' review. Per RECIST 1.1, CR or PR was confirmed by repeated radiographic assessment no less than 4 weeks from the first documented response. If site-assessed PD was verified by the central imaging vendor, the site could elect to continue treatment, repeat imaging ≥4 weeks later and assess tumor response or confirmed progression per irRECIST. The percentage of participants who experienced a CR or PR per RECIST 1.1 or irCR or irPR per irRECIST as assessed by central radiologists' review was reported for each arm per protocol for first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Percentage of participants | 0.0 [0.0 to 23.2] | 23.1 [5.0 to 53.8] | 20.0 [4.3 to 48.1]

12. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Central Radiologists' Review
Description: For participants who demonstrated a confirmed CR (disappearance of all lesions) or confirmed PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by central radiologists' review, DOR was defined as the time from first documented evidence of a CR or PR until disease progression or death. RECIST 1.1 has been modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The DOR per RECIST 1.1 as assessed by central radiologists' review for all participants who experienced a confirmed CR or PR was reported for each arm per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment, had measurable disease at baseline as assessed by central radiology review, and who demonstrated a confirmed response (CR or PR). No participants in the Pembrolizumab 2 mg/kg group were eligible for this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 0 | 3 | 3
Months |  | 6.28 [2.00 to 6.28] | 4.1 [2.00 to 4.11]

13. Secondary Outcome: DOR Per irRECIST as Assessed by Central Radiologists' Review
Description: For participants who demonstrated confirmed CR (disappearance of all target lesions and non-target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 or CR or PR after a single PD, DOR was defined as the time from the first documented CR or PR, or irCR or irPR, until an immune-related progressive disease (irPD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per irRECIST, irPD was defined as after a single PD, ≥20% increase in the sum of diameters of target lesions, or unequivocal worsening of non-target lesions or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. DOR per irRECIST assessed by central radiologists' review for all participants with confirmed CR or PR or irCR or irPR was reported for each arm per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment, had measurable disease at baseline as assessed by central radiology review, and who demonstrated a confirmed response (iCR or iPR). No participants in the Pembrolizumab 2 mg/kg group were eligible for this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 0 | 3 | 3
Months |  | NA [NA to NA] — NA=The median of DOR and the lower and upper ranges of DOR were not reached (no progressive disease by time of last disease assessment). | NA [NA to NA] — NA=The median of DOR and the lower and upper ranges of DOR were not reached (no progressive disease by time of last disease assessment).

14. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by Central Radiologists' Review
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as either a 20% increase from nadir in target lesions, unequivocal progression of nontarget lesions, or the appearance of new lesions. PFS per RECIST 1.1 as assessed by central radiologists' review was reported for each arm per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Months | 2.1 [2.0 to 4.2] | 2.7 [2.1 to 8.2] | 2.1 [1.3 to 6.4]

15. Secondary Outcome: PFS Per irRECIST as Assessed by Central Radiologists' Review
Description: PFS was defined as the time from randomization to the first documented immune-based confirmed progressive disease (iCPD) or death due to any cause, whichever occurred first. Per iRECIST, iCPD is defined as worsening of any existing cause of progression, or the appearance of any other cause of progression, relative to the initial appearance of progressive disease by RECIST 1.1. PFS per irRECIST as assessed by central radiologists' review is reported for each arm per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Months | 2.2 [2.0 to 4.4] | 6.2 [2.1 to NA] — NA=The upper limit of the PFS 95% confidence interval (CI) was not reached by the time of the 19-Sept-2017 data cut-off. | 6.4 [1.3 to NA] — NA=The upper limit of the PFS 95% confidence interval (CI) was not reached by the time of the 19-Sept-2017 data cut-off.

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was reported for each arm using a 19-Sept-2017 data cut-off date per protocol for the first course of treatment.
Time Frame: Up to ~13 months (through Final Analysis database cut-off date of 19-Sept-2017)
Population: All randomized participants that received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Pembrolizumab 200 mg Fixed Dose
Number analyzed (Participants) | 14 | 13 | 15
Months | NA [4.4 to NA] — NA=The median of OS and the upper limit of the OS 95% CI were not reached by the time of the 19-Sept-2017 data cut-off. | 9.4 [6.2 to NA] — NA=The upper limit of the OS 95% CI was not reached by the time of the 19-Sept-2017 data cut-off. | NA [1.3 to NA] — NA=The median of OS and the upper limit of the OS 95% CI were not reached by the time of the 19-Sept-2017 data cut-off.

ADVERSE EVENTS:
Time Frame: Up to ~65 months (through End of Trial database cut-off date of 31-Dec-2021)
Description: All-Cause Mortality was reported according to treatment course for all randomized participants.
  Serious and Other AEs were reported according to treatment course for all randomized participants who received ≥1 dose of study treatment. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab 2 mg/kg First Course: Participants received pembrolizumab 2 mg/kg administered IV Q3W for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days
- Pembrolizumab 10 mg/kg First Course: Participants received pembrolizumab 10 mg/kg administered IV Q3W for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days.
- Pembrolizumab 200 mg Fixed Dose First Course: Participants received pembrolizumab 200 mg fixed dose administered IV Q3W for up to 35 administrations. Cycle 1 was 28 days and subsequent cycles were 21 days.
- Pembrolizumab 2 mg/kg Second Course: Eligible participants who stopped the initial course of pembrolizumab (2 mg/kg administered IV Q3W for up to 35 administrations) with Stable Disease (SD) or better but progressed after discontinuation initiated a second course of pembrolizumab at the same dose per the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Pembrolizumab 2 mg/kg First Course | Pembrolizumab 10 mg/kg First Course | Pembrolizumab 200 mg Fixed Dose First Course | Pembrolizumab 2 mg/kg Second Course
All-Cause Mortality (participants affected / at risk) | 11/14 | 12/15 | 13/15 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/13 | 3/15 | 0/1
Other Adverse Events (participants affected / at risk) | 14/14 | 13/13 | 14/15 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 2 mg/kg First Course (N=14) | Pembrolizumab 10 mg/kg First Course (N=13) | Pembrolizumab 200 mg Fixed Dose First Course (N=15) | Pembrolizumab 2 mg/kg Second Course (N=1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 2 mg/kg First Course (N=14) | Pembrolizumab 10 mg/kg First Course (N=13) | Pembrolizumab 200 mg Fixed Dose First Course (N=15) | Pembrolizumab 2 mg/kg Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (7) | 4 (6) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 3 (3) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (5) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 5 (6) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 4 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (2) | 4 (5) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02835690/Prot_SAP_001.pdf